CLINICAL TRIAL: NCT00805142
Title: Phase II Study of JNS024PR in Cancer Pain Patients
Brief Title: Phase 2 Study of Tapentadol Prolonged Release in Cancer Pain Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015532; JNS024PR-JPN-C01
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-06

CONDITIONS: Pain; Cancer
Keywords: Pain; Cancer; Tapentadol
MeSH Terms: conditions — Pain; Neoplasms | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opioid-Naive Participants (Tapentadol PR) (Experimental): Opioid-naive participants are defined as those who had moderate to severe cancer pain that is not controlled sufficiently with non-opioid medications. Treatment period comprises of Titration and Maintenance period. Titration period (3-14 days) is duration between start of treatment to day before initial dose in the maintenance period. Treatment will be initiated with tapentadol prolonged release (JNS024PR, PR) 25 milligram (mg) oral tablet twice daily. Dose will be increased or decreased as per Investigator's discretion up to Day 14. Maximum dose limit will be 500 mg per day. Participants will then be assigned to the treatment in the maintenance period (15-19 days). The maintenance period is duration between the first dose and the final assessment in the maintenance period. Participants will receive tapentadol PR oral tablet twice daily for 5 days at the same dose used on last day of titration period.
  Interventions: Drug: Tapentadol PR
- Opioid-Switch Participants (Tapentadol PR) (Experimental): Opioid-switching participants are defined as those who had moderate to severe cancer pain that is controlled sufficiently with opioid therapy. Treatment period comprises of Titration and Maintenance period. Titration period (3-14 days) is duration between start of treatment to day before initial dose in maintenance period. Initial dose of tapentadol PR is selected according to daily dose of opioid (morphine sustained release [SR] preparation, oxycodone hydrochloride [HCl] SR tablet or fentanyl patch). Equivalent dose of tapentadol PR oral tablet twice daily is given depending on daily dose of opioid at completion of Screening period. Maximum dose limit is 500 mg per day. Participants will then be assigned to treatment in maintenance period (15-19 days). Maintenance period is defined as duration between first dose and final assessment in maintenance period. Participants will receive tapentadol PR oral tablet twice daily for 5 days at same dose used on last day of titration period.
  Interventions: Drug: Tapentadol PR

INTERVENTIONS:
Drug: Tapentadol PR — Tapentadol PR tablets will be administered orally twice daily initiated at dose of 25 mg. Dose will be adjusted as per Investigator's discretion. Maximum dose limit is 500 mg per day. Total duration of treatment is 19 days.
  Other Names: Tapentadol hydrochloride, JNS024

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time; explores what the body does to the drug) of tapentadol prolonged release (JNS024PR, PR) in participants with moderate to severe cancer (abnormal tissue that grows and spreads in the body until it kills) pain.

DETAILED DESCRIPTION:
This is a Phase 2 open-label (all people know the identity of the intervention), multi-centric (conducted in more than one center), non-comparative, optional dose-titration study of tapentadol PR in Japanese participants with cancer pain. This study will consist of Screening period (3 to 7 days), Dose adjustment period (3 to 14 days), Fixed dose period (5 days) and Follow-up period (7 days). Tapentadol PR will be administered orally (taken by mouth; to be swallowed) twice daily before meal. For participants previously using opioids, the initial dose of tapentadol PR will be selected depending on the daily dose of opioid at the completion of Screening period. For opioid-naive (moderate to severe cancer pain that is not controlled adequately with non-opioid medications) participants, the initial dose of tapentadol PR will be 25 milligram (mg) twice daily. Participants will receive the same dose of tapentadol PR for the first 2 days of the dose adjustment period and from Day 3, the dose can be titrated as per the Investigator's discretion up to Day 14. After that participants will receive fixed dose regimen for 5 days at the same dose as that used at the end of the dose adjustment period. Efficacy will primarily be evaluated by sustained pain control for the 5 day fixed dose phase. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Opioid switching participants should meet the following criteria from a to c: a) Participants with cancer pain b) previously were on opioid medications (morphine sustained release preparations [120 milligram per day {mg/day} or less], oxycodone hydrochloride sustained release tablets [80 mg/day or less], fentanyl transdermal [through the skin] application system [4.2 mg or less]) c) had achieved adequate pain control with opioid therapy
* Opioid naive participants should meet the following criteria from a to b: a) Participants with cancer pain b) should not have received any pain control therapy with opioids (excluding narcotic antagonist analgesics [drug used to control pain])
* Definite diagnosis of any type of cancer, which has been notified to the participant
* Participants who can be hospitalized during the treatment period
* Participant who can record 11 point Numerical Rating Scale (NRS) and 100 millimeter (mm) Visual Analog Scale (VAS) scores appropriately throughout the study

Exclusion Criteria:

* Participants with bradyarrhythmia (slow, irregular heartbeats)
* History of mild or moderate traumatic (causing damage, like a toll used to crush tissue) encephalopathy, cerebral (having to do with the cerebrum) infarction (death of tissue because of lack of blood supply) or transient ischemic (decreased oxygen in a tissue [usually because of decreased blood flow]) attack within 1 year before informed consent
* Previous or concurrent epilepsy (seizure disorder) or convulsive diseases accompanied by disturbance of consciousness
* Previous or concurrent alcohol dependence or narcotic abuse
* History of active hepatitis (inflammation of the liver) B or C within 3 months before informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (21):
- Japan (21):
  - Chiba
  - Chikushino-shi
  - Fukuoka
  - Himeji
  - Hirosaki
  - Ichinomiya
  - Ikeda
  - Iwakuni
  - Kobe
  - Kochi
  - Kyoto
  - Nishinomiya
  - Ohta
  - Osaka
  - Sapporo
  - Sasebo
  - Shizuoka
  - Sonogishukugō
  - Tokyo
  - Toyonaka
  - Utsunomiya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 95 participants signed the informed consent form, of which 78 participants were enrolled in the study.
Groups:
- Opioid-Naive Participants (Tapentadol PR): Opioid-naive participants were defined as those who had moderate to severe cancer pain that was not controlled sufficiently with non-opioid medications. Treatment period comprises of Titration and Maintenance period. Titration period (3-14 days) was duration between start of treatment to day before initial dose in the maintenance period. Treatment was initiated with tapentadol prolonged release (JNS024PR, PR) 25 milligram (mg) oral tablet twice daily. Dose was increased or decreased as per Investigator's discretion up to Day 14. Maximum dose limit was 500 mg per day. Participants were then assigned to the treatment in the maintenance period (15-19 days). The maintenance period was duration between the first dose and the final assessment in the maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at the same dose used on last day of titration period.
- Opioid-Switch Participants (Tapentadol PR): Opioid-switching participants were defined as those who had moderate to severe cancer pain that was controlled sufficiently with opioid therapies. Treatment period comprises of Titration and Maintenance period. Titration period (3-14 days) was duration between start of treatment to day before initial dose in maintenance period. Initial dose of tapentadol PR was selected according to daily dose of opioid (morphine sustained release [SR] preparation, oxycodone hydrochloride [HCl] SR tablet or fentanyl patch). Equivalent dose of tapentadol PR oral tablet twice daily given depending on daily dose of opioid at completion of Screening period. Maximum dose limit was 500 mg per day. Participants were then assigned to treatment in maintenance period (15-19 days). Maintenance period was defined as duration between first dose and final assessment in maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at same dose used on last day of titration period.
Period: Titration Period
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Started | 36 | 42
Completed | 30 | 32
Not Completed | 6 | 10
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Disease Progression | 2 | 1
Not completed — Withdrawal of consent | 0 | 1
Not completed — Other | 0 | 3
Period: Maintenance Period
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Started | 30 | 32
Completed | 30 | 30
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Opioid-Naive Participants (Tapentadol PR): Opioid-naive participants were defined as those who had moderate to severe cancer pain that was not controlled sufficiently with non-opioid medications. Treatment period comprises of Titration and Maintenance period. Titration period (3-14 days) was duration between start of treatment to day before initial dose in the maintenance period. Treatment was initiated with tapentadol prolonged release (PR) 25 milligram (mg) oral tablet twice daily. Dose was increased or decreased as per Investigator's discretion up to Day 14. Maximum dose limit was 500 mg per day. Participants were then assigned to the treatment in the maintenance period (15-19 days). The maintenance period was duration between the first dose and the final assessment in the maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at the same dose used on last day of titration period.
- Opioid-Switch Participants (Tapentadol PR): Opioid-switching participants were defined as those who had moderate to severe cancer pain that was controlled sufficiently with opioid therapies. Treatment period comprised of Titration and Maintenance period. Titration period (3-14 days) was duration between start of treatment to day before initial dose in maintenance period. Initial dose of tapentadol PR was selected according to daily dose of opioid (morphine sustained release [SR] preparation, oxycodone hydrochloride [HCl] SR tablet or fentanyl patch). Equivalent dose of tapentadol PR oral tablet twice daily given depending on daily dose of opioid at completion of Screening period. Maximum dose limit was 500 mg per day. Participants were then assigned to treatment in maintenance period (15-19 days). Maintenance period was defined as duration between first dose and final assessment in maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at same dose used on last day of titration period.
- Total: Total of all reporting groups
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR) | Total
Number analyzed (Participants) | 30 | 36 | 66
Age Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 78 participants, Baseline characteristic (Age) was available for only 66 participants who were included in per protocol (PP) population.
  years | 71.7 (9.97) | 70.0 (8.44) | 70.7 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 78 participants, Baseline characteristic (Gender) was available for only 66 participants who were included in PP population
  Participants
    Female | 10 | 14 | 24
    Male | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Pain Control for 5 Day Fixed Dose Phase
Description: Percentage of participants with sustained pain control for 5 day fixed dose phase were the participants who completed 5 day maintenance period, whose mean Numerical Rating Scale (NRS) score during the fixed dose phase and which was assessed immediately before giving each dose was less than 4 and the number of rescue doses per day for fixed dose phase was 2 or less. Pain intensity scores were recorded 0 to 30 minutes before dose on 11 point NRS where 0 = no pain and 10 = severest pain imaginable.
Time Frame: Day 15 up to Day 19
Population: Per protocol set (PPS) included all participants enrolled excluding those with a major protocol violation. Here 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Opioid-Naive Participants Maintenance Period (Tapentadol PR): Opioid-naive participants were defined as those who had moderate to severe cancer pain that was not controlled adequately with non-opioid medications. The maintenance period (15-19 days) was the duration between the first dose and the final assessment in the maintenance period. Participants received tapentadol prolonged release (PR) oral tablet twice daily for 5 days at the same dose used on last day of titration period.
- Opioid-Switch Participants Maintenance Period (Tapentadol PR): Opioid-switching participants were defined as those who had moderate to severe cancer pain that was controlled sufficiently with opioid therapies. The maintenance period (15-19 days) was defined as the duration between the first dose and the final assessment in the maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at the same dose used on last day of titration period.
Arm/Group | Opioid-Naive Participants Maintenance Period (Tapentadol PR) | Opioid-Switch Participants Maintenance Period (Tapentadol PR)
Number analyzed (Participants) | 29 | 28
percentage of participants | 89.7 [72.6 to 97.8] | 92.9 [76.5 to 99.1]

2. Secondary Outcome: Percentage of Participants Who Achieve Dose Adjustment
Description: Percentage of participants who achieved dose adjustment included those participants whose dose was adjusted during the titration period period and entered the fixed dose maintenance period. Titration period (3-14 days) was the duration between start of treatment to the day before the initial dose in the maintenance period. Maintenance period (15-19 days) was the duration between the first dose and the final assessment in the maintenance period.
Time Frame: Day 3 up to Day 14
Population: The PPS included all participants enrolled excluding those with a major protocol violation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Opioid-Naive Participants Titration Period (Tapentadol PR): Opioid-naive participants were defined as those who had moderate to severe cancer pain that was not controlled sufficiently with non-opioid medications. Titration period (3-14 days) was the duration between start of treatment to the day before the initial dose in the maintenance period. Treatment was initiated with tapentadol PR 25 mg oral tablet twice daily. Dose was increased or decreased as per Investigator's discretion up to Day 14. Maximum dose limit was 500 mg per day.
- Opioid-Switch Participants Titration Period (Tapentadol PR): Opioid-switching participants were defined as those who had moderate to severe cancer pain that was controlled sufficiently with opioid therapies. Titration period (3-14 days) was the duration between start of treatment to the day before the initial dose in the maintenance period. Initial dose of tapentadol PR was selected according to the daily dose of opioid (morphine sustained release (SR) preparation, oxycodone hydrochloride (HCl) SR tablet or fentanyl patch). Equivalent dose of the tapentadol PR oral tablet twice daily given depending on daily dose of opioid at completion of Screening period. Maximum dose limit was 500 mg per day.
Arm/Group | Opioid-Naive Participants Titration Period (Tapentadol PR) | Opioid-Switch Participants Titration Period (Tapentadol PR)
Number analyzed (Participants) | 30 | 36
percentage of participants | 93.3 [77.9 to 99.2] | 80.6 [64.0 to 91.8]

3. Secondary Outcome: Pain Assessment Using 24-hour Numerical Rating Scores (NRS) Scale
Description: Pain intensity scores were measured on 11 point NRS, where 0 = no pain and 10 = severest pain imaginable. The pain intensity at Baseline was the average of scores on two consecutive morning doses (Day -1 and Day 0) and on Day 20 only a single observation was recorded.
Time Frame: Baseline (Average of Day -1 and Day 0 morning scores), Day 20
Population: The PPS included all participants enrolled excluding those with a major protocol violation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Number analyzed (Participants) | 30 | 36
units on a scale
  Baseline | 4.9 (1.40) | 1.3 (1.30)
  Day 20 | 2.4 (1.22) | 1.7 (1.74)

4. Secondary Outcome: Pain Assessment Using Visual Analog Scale (VAS) Score
Description: Pain VAS assesses the pain intensity experienced by the participant on a 100 millimeter (mm) VAS, where responses range from a response of no pain (score of 0 mm) to severest pain imaginable (score of 100 mm). The participant indicated the pain by marking the applicable place with slash (/) and the investigator then measured the length from left edge to the slash.
Time Frame: Baseline and Day 19
Population: The PPS included all participants enrolled excluding those with a major protocol violation. Missing values were imputed using last observed carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Number analyzed (Participants) | 30 | 36
mm
  Baseline | 44.34 (12.870) | 10.71 (11.623)
  Day 19 | 20.33 (10.874) | 10.30 (11.098)

5. Secondary Outcome: Rescue Doses
Description: The immediate release (IR) oral opioids were used as rescue doses in the participants with lack of efficacy or to have relief from severe pain. In case of opioid-switching participants rescue doses were continued without any change in the preceding doses or the type throughout the study. The IR morphine HCl was used as the rescue dose for opioid-naive participants. The upper limit of rescue doses was specified for each daily dose of tapentadol PR. There was no change in the dose of rescue medication during maintenance period for opioid-naive participants.
Time Frame: Day 12, 13, 14, 15, 16, 17, 18 and 19
Population: The PPS included all participants enrolled excluding those with a major protocol violation. Here 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Number analyzed (Participants) | 29 | 28
mg per day
  Day 12 | 0.34 (1.289) | 1.07 (2.562)
  Day 13 | 0.52 (1.550) | 1.16 (2.380)
  Day 14 | 1.03 (2.061) | 1.61 (3.400)
  Day 15 | 1.21 (3.178) | 2.05 (4.503)
  Day 16 | 1.72 (3.348) | 1.21 (2.795)
  Day 17 | 1.72 (3.605) | 1.56 (3.513)
  Day 18 | 0.86 (1.922) | 2.32 (5.639)
  Day 19 | 1.03 (2.061) | 1.96 (4.200)

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Because of Any Adverse Event (AE) or Lack of Efficacy
Description: The AE is an undesirable or unwanted consequence that occurred during the course of the clinical trial, but not necessarily because of study drug.The AEs included the onset of new symptoms, worsening of the frequency or severity of the symptom compared with Baseline, and abnormal findings including abnormal laboratory test values in the diagnostic examination. The participants who discontinued because of lack of efficacy were those in which satisfactory analgesia was not maintained.
Time Frame: Baseline up to 7 days after last dose of study treatment
Population: The PPS included all participants enrolled excluding those with a major protocol violation.
Measure: Number; unit: participants
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Number analyzed (Participants) | 30 | 36
participants
  AEs | 2 | 3
  Lack of efficacy | 0 | 1

7. Secondary Outcome: Sleep Questionnaire Regarding Time to Sleep and Total Time Slept
Description: The sleep questionnaire is a 4-item questionnaire evaluating the condition of the sleep of the participant on the previous night. The participants were asked about the time taken by them to fall asleep previous night after bedtime and the total time they slept during previous night.
Time Frame: Pre-dose (Day 1) and Day 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Opioid-Switch Participants Maintenance Period (Tapentadol PR): Opioid-switching participants were defined as those who had moderate to severe cancer pain that was controlled sufficiently with opioid therapies. Treatment period comprised of Titration and Maintenance period. Titration period (3-14 days) was duration between start of treatment to day before initial dose in maintenance period. Initial dose of tapentadol PR was selected according to daily dose of opioid (morphine sustained release [SR] preparation, oxycodone hydrochloride [HCl] SR tablet or fentanyl patch). Equivalent dose of tapentadol PR oral tablet twice daily given depending on daily dose of opioid at completion of Screening period. Maximum dose limit was 500 mg per day. Participants were then assigned to treatment in maintenance period (15-19 days). Maintenance period was defined as duration between first dose and final assessment in maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at same dose used on last day of titration period.
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants Maintenance Period (Tapentadol PR)
Number analyzed (Participants) | 29 | 28
minutes
  Time to sleep: Pre-dose (Day 1) | 47.10 (44.45) | 63.80 (60.70)
  Time to sleep: Day 20 | 43.10 (39.47) | 56.60 (40.85)
  Total time slept: Pre-dose (Day 1) | 371.70 (119.49) | 390.50 (106.90)
  Total time slept: Day 20 | 418.40 (104.21) | 373.00 (99.40)

8. Secondary Outcome: Sleep Questionnaire Regarding Number of Awakenings
Description: The sleep questionnaire is a 4-item questionnaire evaluating the condition of the sleep of the participant on the previous night . Participants were asked to provide the number of times they awoke at night.
Time Frame: Pre-dose (Day 1) and Day 20
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Number analyzed (Participants) | 29 | 28
awakenings
  Pre-dose (Day 1) | 2.40 (1.70) | 3.40 (2.28)
  Day 20 | 2.20 (1.38) | 3.80 (1.81)

9. Secondary Outcome: Sleep Questionnaire Regarding the Quality of Sleep
Description: The sleep questionnaire is a 4-item questionnaire evaluating the condition of the sleep of the participant on the previous night. Participants rated overall sleep quality on a scale ranging from excellent to very poor.
Time Frame: Pre-dose (Day 1) and Day 20
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Number analyzed (Participants) | 29 | 28
participants
  Excellent: Pre-dose (Day 1) | 1 (3.4) | 0 (0.0)
  Excellent: Day 20 | 4 (13.8) | 2 (7.1)
  Good: Pre-dose (Day 1) | 16 (55.2) | 20 (71.4)
  Good: Day 20 | 17 (58.6) | 18 (64.3)
  Fair: Pre-dose (Day 1) | 0 | 0
  Fair: Day 20 | 8 | 6
  Poor: Pre-dose (Day 1) | 10 | 6
  Poor: Day 20 | 0 | 2
  Very Poor: Pre-dose (Day 1) | 2 | 2
  Very Poor: Day 20 | 0 | 0

10. Secondary Outcome: Patient's Global Impression of Change (PGI-C)
Description: PGI-C is a participant rated instrument to measure participant's change in overall status of general condition including pain on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 19
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Opioid-Naive Participants Maintenance Period (Tapentadol PR): Opioid-naive participants were defined as those who had moderate to severe cancer pain that was not controlled adequately with non-opioid medications. The maintenance period (15-19 days) was the duration between the first dose and the final assessment in the maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at the same dose used on last day of titration period.
- Opioid-Switch Participants Maintenance Period (Tapentadol PR): Opioid-switching participants were defined as those who had moderate to severe cancer pain that was controlled sufficiently with opioid therapies. The maintenance period (15-19 days) was defined as duration between the first dose and the final assessment in the maintenance period. Participants received tapentadol PR oral tablet twice daily for 5 days at the same dose used on last day of titration period.
Arm/Group | Opioid-Naive Participants Maintenance Period (Tapentadol PR) | Opioid-Switch Participants Maintenance Period (Tapentadol PR)
Number analyzed (Participants) | 29 | 28
participants
  Very much improved | 1 (3.4) | 0 (0.0)
  Improved | 13 (44.8) | 1 (3.6)
  Minimally improved | 10 (34.5) | 6 (21.4)
  No change | 5 (17.2) | 15 (53.6)
  Minimally worse | 0 (0.0) | 6 (21.4)
  Worse | 0 (0.0) | 0 (0.0)
  Very much worse | 0 (0.0) | 0 (0.0)

ADVERSE EVENTS:
Time Frame: Baseline up to 7 days after last dose of study treatment
Description: Safety Population consisted of participants who received at least one dose of study medication.
Arm/Group | Opioid-Naive Participants (Tapentadol PR) | Opioid-Switch Participants (Tapentadol PR)
Serious Adverse Events (participants affected / at risk) | 5/36 | 3/42
Other Adverse Events (participants affected / at risk) | 33/36 | 29/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid-Naive Participants (Tapentadol PR) (N=36) | Opioid-Switch Participants (Tapentadol PR) (N=42)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid-Naive Participants (Tapentadol PR) (N=36) | Opioid-Switch Participants (Tapentadol PR) (N=42)
Blood pressure increased (Investigations) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Pyrexia (General disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 19 | 11
Vomiting (Gastrointestinal disorders) | 17 | 6
Constipation (Gastrointestinal disorders) | 15 | 4
Somnolence (Nervous system disorders) | 12 | 5
Anorexia (Metabolism and nutrition disorders) | 4 | 3
White blood cell count decreased (Investigations) | 2 | 5
Dizziness (Nervous system disorders) | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
White blood cell count increased (Investigations) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.